CLINICAL TRIAL: NCT03806465
Title: An Evaluation of the Pilot Implementation of RTS,S/AS01 Through Routine Health Systems in Moderate to High Malaria Transmission Settings in Africa
Brief Title: Malaria Vaccine Pilot Evaluation
Acronym: MVPE
Status: Completed | Type: Observational
Sponsor: Rafiq OKINE (Other)
Responsible Party: Sponsor-Investigator, Rafiq OKINE, Medical Officer, World Health Organization
Organization: World Health Organization (Other)
Other Study IDs: RTSS MVPE
Record Dates: First submitted 2018-12-14; First posted 2019-01-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Malaria,Falciparum; Feasibility; Safety; Mortality
Keywords: Vaccine; Malaria; Africa; Child
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Feasibility survey: These will be children living in the vaccinating and in non-vaccinating areas aged less than 5 years of age. For the midline household survey, this would be restricted to children aged 12-23 months of age.
  Interventions: Other: Feasibility survey
- Sentinel hospital surveillance: These will be children living in the vaccinating and in non-vaccinating areas aged less than 5 years of age who are hospitalized in the 18 sentinel hospitals.
  Interventions: Other: Sentinel hospital surveillance
- Community mortality surveillance: These will be children whose deaths are reported in the vaccinating and in non-vaccinating areas aged less than 5 years of age .
  Interventions: Other: Community mortality surveillance

INTERVENTIONS:
Other: Feasibility survey — A survey questionnaire will be administered at each household. At the baseline household survey, each child aged less than 5 years will be tested for malaria using a rapid malaria test.
  Groups: Feasibility survey
Other: Sentinel hospital surveillance — Cerebrospinal samples will be collected from all children hospitalised and suspected of having meningitis.
  Groups: Sentinel hospital surveillance
Other: Community mortality surveillance — A verbal autopsy will be performed
  Groups: Community mortality surveillance

SUMMARY:
The RTS,S/AS01 malaria vaccine is being introduced sub-nationally in phased pilot introductions through the EPI programmes in Malawi Ghana and Kenya. Vaccine introduction is by the respective MoH in selected areas randomly assigned to receive the vaccine at the beginning of the pilots. In the context of this programmatic activity, the Malaria Vaccine Pilot Evaluation (MVPE) registered here as observational evaluations during early vaccine introduction, include a series of 3 household surveys, and sentinel hospital and community mortality surveillance, building on routine systems.

These observational evaluations will measure:

1. The programmatic feasibility of delivering a 4 dose schedule;
2. Safety in routine use, with focus on cerebral malaria and meningitis;
3. The impact of the malaria vaccine in routine use on severe malaria and all-cause mortality

DETAILED DESCRIPTION:
An evaluation of the pilot implementation of RTS,S/AS01 through routine health systems in moderate to high malaria transmission settings in Ghana, Kenya and Malawi. In the context of the new vaccine introduction, the Ministries of Health in the three countries will introduce the malaria vaccine (RTS,S/AS01) in a phased fashion (with some areas introducing the malaria vaccine first and the latter half, after the evaluation period) building on the national immunization programmes which routinely deliver vaccines and expanding the schedule of their routine EPI contacts.

The evaluation of the pilot implementation will run for a total of about 46 months in each country. This will focus on the three main primary objectives of feasibility, safety and impact. The pilot implementation assumes that a total of 46-60 clusters will be identified per country, evenly split between implementation and comparison areas, with each cluster contributing approximately 4,000 children per year to the evaluation of RTS,S/AS01. Hence a total of approximately 120,000 children will receive the RTS,S vaccine in each country in each year. Evaluation data will be collected in the following ways.

COMMUNITY BASED MORTALITY SURVEILLANCE

Community based mortality surveillance will be established across the pilot evaluation areas to enable the evaluation of the impact of the malaria vaccine on all-cause mortality. This will use a network of Village Reporters (VR) to document all deaths among children aged up to 48 months in the implementation and comparison areas. Once the death is notified, a standardized, WHO-approved Verbal Autopsy (VA) will be performed, according to WHO guidelines and locally acceptable practices. The VA will focus is on confirming death, age and vaccination status. The total number of clusters per country is expected to range from 46-60. Assuming 4,000 children born per cluster per year, 30 months of vaccination and a total follow-up of 44 months, each cluster will contribute 23,134 person years at risk (pyar), allowing for 1% mortality in the first month of life, and 0.08% mortality for every month after the first month. This equates to a mortality risk of 22.2 per 1000 for children aged 5 to 36 months. A mortality risk of 21 per 1,000 equates to a rate, over 2.5 years, of 8.489455 per 1,000 pyar. Based on a minimum mortality rate of 8.5 per 1000 pyar, 23 clusters in each arm, each with an annual birth cohort of approximately 4,000 subjects, would have 80% power to detect, at the 5% significance level, a decrease of at least 10% in overall mortality in each country.

With this mortality risk, the pilot evaluation it is estimated to have approximately 80% power to detect an interaction between gender and treatment of 1.15 (i.e an increased risk of mortality in girls of 1.035), compared with the 1.9-fold increase in risk among girls receiving RTS,S/AS01 in the RTS,S Phase 3 trial.

FEASIBILITY (CROSS SECTIONAL HOUSEHOLD) SURVEYS)

Three household surveys will be conducted to evaluate the programmatic feasibility to deliver a 4 dose schedule at baseline (before vaccination starts), 18 months and 30 months after start of vaccination.

A sample size of 100 houses per cluster will estimate the cluster-specific coverage of RTS,S/AS01 to within 10% (ie 95% CI from 40 to 60%) using a conservative estimate of 50% coverage and a high response rate above 95% in each cluster. Assuming a design effect of 1.5 between clusters, the overall precision in RTS,S/AS01 and coverage estimates of other vaccines over the pilot programme's implementation and comparison areas will be 2% (ie 95%CI 48% to 52%) in each country. This will result in 15,800 (6,600 in Ghana, 4,600 each in Kenya and Malawi) households included in the surveys. The second household survey may be powered to generate coverage estimates in each arm, rather than in each cluster, to within ±2% of the true value.

SENTINEL HOSPITAL SURVEILLANCE

Four to eight sentinel hospitals will be identified in each country to collect information on a larger scale on the safety of the malaria vaccine in children aged less than 5 years admitted with a focus on cases of cerebral malaria and meningitis. The catchment area of each hospital (approximately a cluster) is expected to have an annual birth cohort of, and provide services for, approximately 4,000 children in the MVPE. Hence a total catchment area of 48,000 children in implementation areas and another 48,000 children in comparison areas will contribute to the hospital-based evaluation of safety across the programme (three countries, Ghana, Kenya and Malawi). This is expected to provide 80% power to detect a 1.7-fold increase in risk of cerebral malaria and 2.6-fold increase in risk of meningitis. Children admitted to the sentinel hospitals in this age group will be assessed for severe malaria and meningitis using a standardised surveillance approach.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-59 months

Exclusion Criteria:

* Children aged less than 1 month or greater than 59 months

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will comprise children aged 1-59 months living in the areas geographically-defined for this evaluation of the RTS,S/AS01 Malaria Vaccine Implementation in three countries (Ghana, Kenya and Malawi) in sub-Saharan Africa.
Sampling Method: Non-Probability Sample
Enrollment: 30124 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The number of deaths of any cause | From 0 to 46 months after vaccination starts
  Number of deaths of any cause in children aged 1-59 months.
Number of children admitted with a diagnosis of probable and confirmed meningitis cases | From 0 to 30 months after vaccination starts
  Number of children with probable and confirmed meningitis A probable case if in a suspected case, the macroscopic aspect of the CSF is turbid, cloudy or purulent; or the CSF leukocyte count is >10 cells/mm3. A confirmed case is if a suspected or probable case is laboratory confirmed by culturing or identifying (i.e. by polymerase chain reaction, immunochromatographic dipstick or latex agglutination) bacterial, viral or other aetiology in the CSF.
Number of children admitted with a diagnosis of cerebral malaria | From 0 to 30 months after vaccination starts
  Cerebral malaria is defined as Severe P. falciparum malaria with coma (Glasgow coma score < 11 in children two years of age or older [≥ 2 years] or Blantyre coma score < 3 in children less than two years of age [(< 2 years]); and If malaria with seizure: coma persisting for > 30 min after the seizure. Other treatable causes of coma should be excluded before diagnosing cerebral malaria (e.g. hypoglycaemia, bacterial meningitis)
Number of children aged 12-23 months who have completed the primary series (the 3 dose regime) of the malaria vaccine | At 18 months after vaccination starts
  Prevalence of children aged 12-23 months who had completed three doses of RTS,S/AS01 at the second household survey
Number of children aged 27-38 months who have completed the 4th dose of the malaria vaccine | At 30 months after vaccination starts
  Prevalence of children aged 27-38 months who had completed four doses of RTS,S/AS01 at the third household survey

SECONDARY OUTCOMES:
Number of deaths in children by gender | From 0 to 46 months after vaccination starts
  Number of deaths in children stratified by gender in children aged 1-59 months
Number of deaths in hospitalised children by gender | From 0 to 46 months after vaccination starts
  Number of deaths in hospitalized children stratified by gender in children aged 1-59 months.
Number of malaria associated deaths in hospitalised children by gender | From 0 to 46 months after vaccination starts
  Number of malaria specific deaths stratified by gender in hospitalized children aged 1-59 months.
Number of children with a diagnosis of severe malaria | From 0 to 30 months after vaccination starts
  Hospital admissions with malaria which meet WHO criteria for a diagnosis of severe malaria.
Number of deaths excluding those attributed to trauma, poisoning and drowning | From 0 to 46 months after vaccination starts
  Number of non traumatic deaths in children aged 1-59 months.
Number of children with a diagnosis of aetiology confirmed meningitis | 30 months after vaccination starts
  Number of hospital admissions which meet WHO criteria for a diagnosis of aetiologically confirmed meningitis admitted to sentinel hospitals
Number of children with a diagnosis of suspected meningitis | From 0 to 30 months after vaccination starts
  Number of hospital admissions which meet WHO criteria for a diagnosis of suspected meningitis admitted to sentinel hospitals
Number of children with a diagnosis of probable meningitis | From 0 to 30 months after vaccination starts
  Number of hospital admissions which meet WHO criteria for a diagnosis of probable meningitis admitted to sentinel hospitals
Number of children with a diagnosis of malaria | From 0 to 30 months after vaccination starts
  Number of hospital admissions which meet WHO criteria for a diagnosis of malaria admitted to sentinel hospitals
Number of children with a non-malaria diagnosis | From 0 to 30 months after vaccination starts
  Number of hospital admissions which do not meet WHO criteria for a diagnosis of malaria admitted to sentinel hospitals
Number of children with a diagnosis of anaemia | From 0 to 30 months after vaccination starts
  Number of hospital admissions which meet WHO criteria for a diagnosis of anaemia admitted to sentinel hospitals . Anaemia is haemoglobin less than 11g/dL.
Number of children who have received all their routine EPI vaccines as recommended by their national immunization schedule | At 18 and 30 months after vaccination starts
  Routine EPI vaccines include all doses of OPV, pentavalent, rotavirus, pneumococcal and measles vaccines
Number of children who have received all the recommended malaria prevention and control measures | At 18 and 30 months after vaccination starts
  Recommended malaria prevention and control measures include insecticide treated bed nets, IPTi and indoor residual spraying.
Number of children who have received all of the other key childhood interventions | At 18 and 30 months after vaccination starts
  Other key childhood interventions include anti-helminth administration (deworming) and Vitamin A supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Don Mathanga, PhD, Principal Investigator — College of Medicine, Malawi; Kwaku Poku Asante, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana; Aaron Samuels, MD, Principal Investigator — CDC-Kenya Malaria Program
Locations (3):
- Kintampo Health Research Centre, Kintampo, Ghana
- CDC Kenya Malaria Programme, Kisumu, Kenya
- College of Medicine, Blantyre, Malawi

REFERENCES:
- [Background] Malaria vaccine: WHO position paper-January 2016. Wkly Epidemiol Rec. 2016 Jan 4;91(4):33-51. No abstract available. English, French. PMID 26829826
- [Background] RTS,S Clinical Trials Partnership. Efficacy and safety of RTS,S/AS01 malaria vaccine with or without a booster dose in infants and children in Africa: final results of a phase 3, individually randomised, controlled trial. Lancet. 2015 Jul 4;386(9988):31-45. doi: 10.1016/S0140-6736(15)60721-8. Epub 2015 Apr 23. PMID 25913272
- [Derived] Hoyt J, Okello G, Bange T, Kariuki S, Jalloh MF, Webster J, Hill J. RTS,S/AS01 malaria vaccine pilot implementation in western Kenya: a qualitative longitudinal study to understand immunisation barriers and optimise uptake. BMC Public Health. 2023 Nov 18;23(1):2283. doi: 10.1186/s12889-023-17194-2. PMID 37980467
- See also: Key milestones in the development of the Malaria Vaccine Implementation Programme (MVIP): from pilot recommendation to vaccine introduction — https://www.who.int/docs/default-source/immunization/mvip/mvip-milestones-to-programme-development-final.pdf?Status=Temp&sfvrsn=14768db0_2

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT03806465/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT03806465/SAP_002.pdf